CLINICAL TRIAL: NCT03671798
Title: Establish a National Registry to Search for the Risk Factors, Etiology, and Neurodegenerative Progression of REM Sleep Behavior Disorder
Brief Title: Establish a National Registry of REM Sleep Behavior Disorder
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Zhang Jihui, Assistant Professor, Chinese University of Hong Kong
Other Study IDs: 2014.445
Record Dates: First submitted 2018-08-30; First posted 2018-09-14 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-08

CONDITIONS: REM Sleep Behavior Disorder
MeSH Terms: conditions — REM Sleep Behavior Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — TFT, Vitamin B12, Folate, CBC, Fasting Glucose, LFT, RFT, CRP, Fasting lipid, Iron profile, Phosphate, Calcium, Neurosteroid, Genetic analysis

GROUPS / COHORTS (2):
- REM sleep behavior disorder (RBD): Diagnosis of RBD according to ICSD-3: 1) Sleep talking or complex movement during sleep. 2) Such movement was recorded by video PSG (AV-PSG) during REM sleep or according to history the movements were occurred during REM. 3) REM sleep without atonia (RWA) during PSG monitoring. 4) This abnormal phenomenon cannot be explained by other sleep disorder, psychiatric disease, drug or substance abuse.
- Controls: Subjects with 1) No RBD symptoms and PSG characteristics. 2) No neurological symptoms or diseases, MRI scan will be employed to exclude brain pathology. 3) No narcolepsy or hypersomnia, ruled out by multiple sleep latency test. 4) No history of mental illnesses or use of antidepressants

SUMMARY:
In this proposed study, the investigators aim to build up a large cohort of Rapid eye movement sleep behavior disorder (RBD) to study the etiology and risk factors of neurodegeneration.

DETAILED DESCRIPTION:
REM sleep behavior disorder (RBD) is a parasomnia characterized by abnormal behavioral manifestations during REM sleep. Accumulating evidence suggests that RBD is implicated as an integral part of disease progress of α-synucleinopathy neurodegeneration, such as Parkinson's disease (PD) and dementia with Lewy bodies.Previous studies have identified a series of neurocognitive, autonomic, clinical and neurobiological markers for neurodegeneration in iRBD, such as olfactory dysfunction, color vision deficit, autonomic dysfunction, tonic EMG activity during REM sleep, and psychiatric disorder. However, the prevalence rate of RBD was relatively low and most of the RBD studies only have 100 or below cases. and there might be ethic differences in RBD which indicates that the findings from western countries might not be applicable to Chinese. In these regards, the investigators aimed to build up a large cohort of Rapid eye movement sleep behavior disorder (RBD) to study the etiology and risk factors of neurodegeneration.

ELIGIBILITY:
Inclusion Criteria:

Case: According to the ICSD-3 for the diagnosis of RBD

1. Sleep talking or complex movement during sleep;
2. Such movement was recorded by video PSG (AV-PSG) during REM sleep or according to history the movements were occurred during REM;
3. REM sleep without atonia (RWA) during PSG monitoring;
4. This abnormal phenomenon cannot be explained by other sleep disorder, psychiatric disease, drug or substance abuse.

Control: Age and gender matched with consent

1. No RBD symptoms and PSG characteristics;
2. No neurological symptoms or diseases, MRI scan will be employed to exclude brain pathology;
3. No narcolepsy or hypersomnia, ruled out by multiple sleep latency test;
4. No history of mental illnesses or use of antidepressants.

Exclusion Criteria:

1. Subjects who refused to join the cohort.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from psychiatry outpatient clinics, Prince of Wales Hospital and 11 collaborated sites in mainland China.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2014-10; Primary Completion 2022-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Risk factors for neurodegenerative diseases in rapid eye movement sleep behavior disorder. | 1 hour
  Risk factors for neurodegenerative diseases were investigated in rapid eye movement sleep behavior disorder by questionnaires, including general information, life history, occupational history and family history.
Changes of neurocognitive biomarkers for neurodegenerative diseases in rapid eye movement sleep behavior disorder. | Baseline and biennial follow-up, up to 20 years
  Based on the large cohort of RBD, the investigators aim to study the etiology and the progression of neurocognitive biomarkers for neurodegenerative diseases in rapid eye movement sleep behavior disorder by clinical assessment, including MoCA, olfactory dysfunction, color vision deficit and so on.
Changes of autonomic dysfunctions for neurodegenerative diseases in rapid eye movement sleep behavior disorder. | Baseline and biennial follow-up, up to 20 years
  Autonomic dysfunctions are also biomarkers for neurodegenerative diseases, the investigators aim to observe the changes of autonomic dysfunctions, including constipation, orthostatic hypotension and so on.
Changes of REM-related EMG activity (REMREEA) and motor activity in rapid eye movement sleep behavior disorder. | Baseline and biennial follow-up, up to 20 years
  The percentage of REM-related EMG activity (REMREEA) is the most reliable and valid marker in differentiating patients with RBD from normal controls. Both REMREEA and significant motor activity were recorded by video-polysomnography in rapid eye movement sleep behavior disorder.

CONTACTS AND LOCATIONS:
Overall Officials: Jihui Zhang, PhD, Principal Investigator — Chinese University of Hong Kong; Yun Kwok Wing, MBChB, Study Director — Chinese University of Hong Kong
Locations (1):
- Department of psychiatry, Faculty of Medicine, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided
Researcher in other sleep centers are also conducting similar study, there may be a plan for further collaboration on sharing the database